CLINICAL TRIAL: NCT00831363
Title: Minimal Invasive Versus Traditional Transgluteal Approach in Total Hip Arthroplasty: a Comparative Gait Analysis
Status: Completed | Type: Observational
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Other Study IDs: GA-0001-MP
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Total Hip Arthroplasty
Keywords: gait analysis; minimal invasive approach; transgluteal approach; THA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: minimal invasive approach
  Interventions: Procedure: minimally invasive total hip arthroplasty
- 2: traditional transgluteal approach
  Interventions: Procedure: standard approach total hip arthroplasty

INTERVENTIONS:
Procedure: minimally invasive total hip arthroplasty — minimally invasive total hip arthroplasty
  Groups: 1
Procedure: standard approach total hip arthroplasty — standard Hardinge approach/traditional transgluteal approach
  Groups: 2

SUMMARY:
The hypothesis for the present study was that patients receiving a minimally invasive total hip arthroplasty will show a faster improvement on walking ability and mobilization in the immediate postoperative period compared to patients with the standard Hardinge approach. Therefore, the main goal was to evaluate the differences in early rehabilitation of these two different surgical approaches by gait analysis and electromyographical examination as objective methods.

ELIGIBILITY:
Inclusion Criteria:

* unilateral osteoarthritis of the hip
* BMI below 30

Exclusion Criteria:

* previous surgery on the evaluated hip,
* previous arthroplasties on other joints,
* a leg length discrepancy of more than 0.5cm,
* rheumatoid osteoarthritis
* decreased mobility due to non joint related factors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Hospital Speising, Vienna, Austria